CLINICAL TRIAL: NCT03178370
Title: Autonomic and Enteric Profiling in Relation to Body Weight
Brief Title: Autonomic and Enteric Profiling
Status: Completed | Type: Observational
Sponsor: University of Louisville (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Thomas Abell, Professor, University of Louisville
Other Study IDs: 13.0890; 5U01DK074007-12 (NIH)
Record Dates: First submitted 2017-05-30; First posted 2017-06-06 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Gastroparesis
Keywords: Gastroparesis; Nausea and Vomiting; Abdominal Pain; Gastric Emptying; Electrophysiology; Hormones; Inflammation; Enteric Nervous System; Autonomic Nervous System
MeSH Terms: conditions — Gastroparesis; Nausea; Vomiting; Abdominal Pain; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Diabetic Gastroparesis
  Interventions: Device: Gastric Electrical Stimulation
- Idiopathic Gastroparesis
  Interventions: Device: Gastric Electrical Stimulation

INTERVENTIONS:
Device: Gastric Electrical Stimulation — Temporary and permanent gastric electrical stimulation

SUMMARY:
Autonomic, inflammatory, enteric, electrophysiologic and hormonal.

DETAILED DESCRIPTION:
Patients were evaluated by two methods in each of five areas: inflammatory, autonomic, enteric, electrophysiologic, and hormonal.

In part one, patients had similar GI Symptoms regardless of baseline gastric emptying or diabetic/non-diabetic status and all patients demonstrated abnormalities in each of the 5 areas studied.

In part two, patients showed early and late effects of electrical stimulation with changes noted in multiple areas, categorized by improvement status.

ELIGIBILITY:
Inclusion Criteria:

1. Willingness to participate in study and sign informed consent.
2. Age 18 or older.
3. Symptoms of gastroparesis for at least 6 months.
4. Refractory or intolerant to antiemetic drugs.
5. Refractory or intolerant to prokinetic drugs.
6. If Diabetic, documentation of medication for diabetes for at least 6 months.
7. No evidence of anatomic obstruction of GI tract. -

Exclusion Criteria:

1. Previous gastric surgery.
2. History or evidence of rumination syndrome, eating disorder of primary psychiatric disorder.
3. No know collagen vascular disease.
4. Inability or unwillingness to participate in the study.
5. Current active gastric stimulation or other gastrointestinal neurostimulation implant or device.
6. Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From 44 consecutive consented patients seen in our clinic, 43 were deemed to be eligible for the study. Those 43 patients were the basis for the baseline evaluation (part one) of this study. Of 43 patients, (description: 15 M, 28 F, mean age 46.3 years; 23 DM, 20 ID), 41 (description: 13 M, 28 F, mean age 45.7 years; 21 DM, 20 ID), finished the temporary phase of gastric electrical stimulation, and 36 (description: 11 M, 25 F, mean age 44.7 years; 18 DM, 18 ID) of those 41 were implanted with permanent GES devices. Of 36 implanted, 30 patients (description: 9 M, 21 F, mean age 43.1 years; 14 DM, 16 ID) were followed at 6 months. The entirety of the GES patients, baseline, temporary and permanent, were the basis for the stimulation portion (part two) of this study.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2014-03-06 (Actual); Primary Completion 2015-12-03 (Actual); Study Completion 2015-12-03 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal symptoms | Change from baseline to 6 days to 6 months
  By standardized symptom scoring

SECONDARY OUTCOMES:
Gastric Emptying Test | baseline, 6 days, 6 months
  By gastric emptying test
Autonomic | Change from baseline to 6 days to 6 months
  By autonomic function
Hormones | Change from baseline to 6 days to 6 months
  By serum measures
Inflammation | Change from baseline to 6 days to 6 months
  By serum measures
Gastric emptying | baseline, 6 days, 6 months
  By radionuclides
Electrophysiology | Change from baseline to 6 days to 6 months
  By Electrogastrogram(EGG)/ Electrogram (EG)
Quality of life by IDIOMS | Change from baseline to 6 days to 6 months
  By standardized scale

IPD SHARING:
Plan to Share IPD: Undecided
No plan in place.

REFERENCES:
- [Derived] Abell TL, Kedar A, Stocker A, Beatty K, McElmurray L, Hughes M, Rashed H, Kennedy W, Wendelschafer-Crabb G, Yang X, Fraig M, Gobejishvili L, Omer E, Miller E, Griswold M, Pinkston C. Pathophysiology of Gastroparesis Syndromes Includes Anatomic and Physiologic Abnormalities. Dig Dis Sci. 2021 Apr;66(4):1127-1141. doi: 10.1007/s10620-020-06259-6. Epub 2020 Apr 23. PMID 32328893
- [Derived] Abell TL, Kedar A, Stocker A, Beatty K, McElmurray L, Hughes M, Rashed H, Kennedy W, Wendelschafer-Crabb G, Yang X, Fraig M, Omer E, Miller E, Griswold M, Pinkston C. Gastroparesis syndromes: Response to electrical stimulation. Neurogastroenterol Motil. 2019 Mar;31(3):e13534. doi: 10.1111/nmo.13534. Epub 2019 Jan 31. PMID 30706646